## Spinal Cord Stimulation to Restore Cough IRB98-00091

NCT number: 00116337

Date of the document: June 27, 2011

Title of Document: Statistical analysis plan

| , |
|---|

## Strategical Analysis Plan

Each patient will serve as their own control; comparisons (e.g. maximum airway and gastric pressure generation and maximum flow rate generation, stimulus amplitude/pressure curves, stimulus frequency/pressure curves, stimulus amplitude/ flow rate curves, stimulus frequency /flow rate curves) will be made at various points in the study. Clinical parameters will be assessed before the study and at several end points following the Reconditioning Phase. Mean changes of each parameter for the entire group and stratified per spinal cord level will be obtained. Statistical analyses will be performed using a repeated measures analysis of variance and Paired t test. A p value of < 0.05 will be taken as indicating statistical significance.

| • |
|---|